CLINICAL TRIAL: NCT07308795
Title: The Ultrasonographic Evaluation of Abdominal Accessory Respiratory Muscle Thickness in Patients With Parkinson's Disease: Correlation With Disease Severity and Expiratory Respiratory Muscle Strength
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayşe Nur Sarıkoç, Assistant Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2025-28
Record Dates: First submitted 2025-12-08; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease (PD); Maximum Inspiratory Pressure; Maximum Expiratory Pressure; Abdominal Accessory Respiratory Muscle Thickness
Keywords: abdominal muscles ultrasonography; parkinson disease; respiratory; MIP; abdominal muscles; respiratory muscles; expiratory muscle strenght; ultrasound; maximum expiratory pressure (MEP)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease (PD): Abdominal Accesory Respiratory Muscles (rectus abdominis, transversus abdominis, and oblique muscles) and MIP(maximum inspiratory pressure) MEP(maximum expiratory pressure) values of the group with Parkinson's diagnosis and Hoehn Yahr Stage 1-2-3 will be measured, a 6-Minute Walk Test will be performed and the results will be noted.
- Control Group: Abdominal Accessory Respiratory Muscles (rectus abdominis, transversus abdominis, and oblique muscles) and MIP (maximum inspiratory muscles) MEP(maximum expiratory muscles) values of age and gender matched healthy values of age and gender matched healthy volunteers without any diagnosis of neuromuscular disease or chest diseases will be measured and the results will be noted.

SUMMARY:
Parkinson's disease is a neurodegenerative disorder characterized by both motor and non-motor symptoms. The involvement of respiratory muscles can lead to impairments in respiratory function in these patients. In this study is to evaluate the thickness of abdominal accessory respiratory muscles using ultrasonography in patients with Parkinson's disease. Additionally, the relationship between disease severity and expiratory respiratory muscle strength will be examined.

The study will include Parkinson's patients at different stages of the disease, with respiratory muscle thickness measured via ultrasonography. The collected data will then be compared with disease severity and expiratory muscle strength.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder characterized by both motor and non-motor symptoms. The involvement of respiratory muscles can lead to impairments in respiratory function in these patients.

This observational, cross sectional study will include Parkinson's patients at different stages of the disease, with respiratory muscle thickness measured via ultrasonography. The collected data will then be compared with disease severity and expiratory muscle strength. In this study is to evaluate the thickness of abdominal accessory respiratory muscles (rectus abdominis, transversus abdominis, and oblique muscles) using ultrasonography in patients with Parkinson's disease. Additionally, the relationship between disease severity and expiratory respiratory muscle strength will be examined. Respiratory muscle strength will be assessed using maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements. Disease severity will be evaluated using standardized clinical scales.

These findings will underscore the importance of evaluating respiratory muscles in Parkinson's disease and may contribute to the development of rehabilitation programs targeting respiratory muscles in the later stages of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Parkinson's disease diagnosis with Modified Hoehn and Yahr stages 1-2-3
* Mini-Mental State Examination (MMSE) score > 23
* Body Mass Index (BMI) < 30

Exclusion Criteria:

* Active smokers
* Individuals with a diagnosis of active chest disease
* Those with hemodynamic instability
* Individuals with unstable vital signs
* Parkinson's patients who cannot be controlled with medical treatment
* Parkinson Plus syndromes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: THE GROUP WITH PARKINSON'S DIAGNOSIS AND HOEHN YAHR STAGE 1-2-3
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Maximal Expiratory Pressure (MEP) Measurement | to be measured only once at the start day 1
  MEP assesses the strength of abdominal and accessory expiratory muscles. During the maneuver, the patient is asked to blow forcefully into the mouthpiece for at least 1.5 seconds, as if inflating a balloon. The pressure generated during rapid expiration is measured by sensors, and after 1.5-2.0 seconds the shutter opens, ending the test. If multiple tests are conducted, the patient rests for at least 1 minute between trials, and a maximum of 3-5 trials are performed. Differences greater than 10 cmH₂O between trials are not accepted. The highest measurement is reported together with the predicted value. The MicroRPM Respiratory Pressure Meter (MicroDirect, USA) will be used.
Maximal Inspiratory Pressure (MIP) Measurement | to be measured only once at the start day 1
  MIP is used to assess the strength of inspiratory respiratory muscles. During the test, the patient is instructed to exhale down to residual volume. MIP is defined as the maximum negative pressure measured during a maximal inspiratory effort performed after reaching residual volume. Measurements will be taken using the MicroRPM Respiratory Pressure Meter (MicroDirect, USA).
Ultrasonographic Assessment of Abdominal Accessory Respiratory Muscles | to be measured only once at the start day 1
  Ultrasound measurements of the rectus abdominis, external oblique, internal oblique, and transversus abdominis muscles will be performed. Measurements will be taken in the supine position with the patient lying on their back, eyes facing upward, arms resting symmetrically beside the trunk, and lower extremities in full knee extension with an intermalleolar distance of 10 cm. Muscle thickness will be recorded at the end of normal expiration and at the end of forced expiration.

OTHER OUTCOMES:
Six Minute Walk Test (6MWT) | to be measured only once at the start day 1
  The 6MWT is performed in a corridor with a flat, firm surface that is at least 30 meters long and marked at 3-meter intervals. Turning points should be indicated with a colored object. Start and finish lines are designated. The patient is asked to walk the longest distance possible within 6 minutes. The distance walked is measured and recorded.
Modified Hoehn and Yahr Staging | to be measured only once at the start day 1
  This scale, developed by Margaret Hoehn and Melvin Yahr in 1967, is used to determine the severity of Parkinson's disease. It evaluates patient functionality, symptom laterality, pattern of involvement, and balance. The scoring ranges from 1 to 5. The Modified Hoehn & Yahr staging system includes additional stages 1.5 and 2.5. As the stage progresses, symptoms become more widespread, balance impairment and functional limitation increase; in the later stages, the patient becomes dependent on assistance or care.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Fizik Tedavi Ve Rehabilitasyon Eğitim Ve Araştirma Hastanesi, Istanbul, BAHÇELİEVLER, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and privacy considerations.